CLINICAL TRIAL: NCT00583505
Title: Emergency/Compassionate Use - Membranous VSD Occluder
Status: No longer available | Type: Expanded Access
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA-008 E/C; G020202
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Membranous; Ventricular; Septal; Defects; VSD
Keywords: membranous; ventricular; septal; defects; VSD

INTERVENTIONS:
Device: Device closure with the AMPLATZER Membranous VSD Occluder — Device closure with the AMPLATZER Membranous VSD Occluder

SUMMARY:
Emergency/Compassionate use of the AMPLATZER Membranous VSD Occluder

ELIGIBILITY:
Inclusion Criteria:

* Emergency/compassionate use for patients not meeting the inclusion critera for the AMPLATZER Membranous VSD clinical trial

Sex: All
Age Groups: Child, Adult, Older Adult